CLINICAL TRIAL: NCT05271929
Title: A Randomised Open-Label Trial of Early, Very High-Titre Convalescent Plasma Therapy in Clinically Vulnerable Individuals With Mild COVID-19
Brief Title: Early High-Titre Convalescent Plasma in Clinically Vulnerable Individuals With Mild COVID-19
Acronym: COVIC-19
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the significant decline in the number of newly diagnosed infections and the difficulties in opening new centers in the outgoing pandemic, recruitment declined. The Data Safety Monitoring Board recommended to stop the trial.
Sponsor: Deutsches Rotes Kreuz DRK-Blutspendedienst Baden-Wurttemberg-Hessen (Other)
Collaborators: NHS Blood and Transplant (Other Government); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVIC-19
Record Dates: First submitted 2022-03-03; First posted 2022-03-09 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current standard of care (Active Comparator): Standard of care therapy may include anti-SARS-CoV-2 specific medication such as, but not limited to:
  * Casirivimab
  * Casirivimab / Imdevimab (REGN-COV2 or Ronapreve)
  * Imdevimab
  * Sotrovimab (Xevudy)
  * Tixagevimab / Cilgavimab (Evusheld)
  * Molnupiravir (MK-4482)
  * Nirmatrevlir / Ritonavir (Paxlovid)
  * Remdesivir
  Centres should ensure that medications used as standard of care are used similarly for patients in both treatment arms.
  Interventions: Other: Current standard of care
- Current standard of care and convalescent plasma (Experimental): Current standard of care and the infusion of two plasma units collected from two different COVID-19 convalescent patients.
  Interventions: Biological: Current standard of care and COVID-19 convalescent and vaccinated plasma

INTERVENTIONS:
Biological: Current standard of care and COVID-19 convalescent and vaccinated plasma — ABO compatible convalescent plasma infused intravenously on study day 1 (as soon as possible after randomisation) and the second on day 1 or day 2. Plasma obtained by apheresis from donors who have recovered from COVID-19 infection (at least 14 days after recovery) and have been vaccinated (at least 3 weeks after first dose of vaccine). A combination of both a SARS-CoV-infection and a SARS-CoV-2 vaccination of the donor is required - irrespective of the sequence of infection and vaccination. As far as the availability of CCP units allows, the two plasma units should have been donated by two different convalescents.
  Arms: Current standard of care and convalescent plasma
Other: Current standard of care — Standard of care therapy may include anti-SARS-CoV-2 specific medication such as, but not limited to:
  * Casirivimab
  * Casirivimab / Imdevimab (REGN-COV2 or Ronapreve)
  * Imdevimab
  * Sotrovimab (Xevudy)
  * Tixagevimab / Cilgavimab (Evusheld)
  * Molnupiravir (MK-4482)
  * Nirmatrevlir / Ritonavir (Paxlovid)
  * Remdesivir
  Centres should ensure that medications used as standard of care are used similarly for patients in both treatment arms.
  Arms: Current standard of care

SUMMARY:
* Research Question: Does convalescent plasma (CCP) collected from donors who have recovered from COVID-19 and who have a very high titre of anti-SARS-CoV-2 antibodies reduce the risk of hospitalisation (for COVID-19) or death in patients with early symptoms of acute COVID-19 who are vulnerable to this disease compared to standard of care?
* Study product: Very high antibody titre COVID-19 convalescent plasma collected more than 15 days after end of symptoms in COVID-19 patients who also had received at least one dose of a SARS-CoV-2 vaccine.
* Methodology: Multicentre, randomised, open-label, adaptive superiority trial: COVID-19 very high neutralizing Ab titre convalescent plasma vs standard care in 2 cohorts of vulnerable patients (cohort 1: elderly (≥ 70 years) and younger with comorbidities, cohort 2: immunosuppressed patients).
* Study phase: Phase 3
* Intervention: Two units of high antibody titre COVID-19 convalescent plasma to individuals randomised to the intervention group, 2 units from 2 different donors, preferably transfused on the same day. Plasma provided by convalescent vaccinated donors with a minimum antibody titre of 1:640 against delta variant (B1.617.2) or antibody concentration >=4.000 BAU/ml in the QuantiVac anti-SARS-CoV-2 IgG ELISA or >=20.000 U/ml in the Elecsys anti-SARS-CoV-2 CLIA
* Randomisation: 1:1 (standard of care + convalescent plasma vs. standard of care) stratified by centre (cohorts 1 and 2)

DETAILED DESCRIPTION:
COVIC-19 is a multicentre international, randomised, open-label adaptive superiority phase III trial to evaluate the efficacy and safety of COVID-19 convalescent plasma in the treatment of COVID-19. It is conducted in a harmonized approach in different countries in Europe.

The study is randomizing adult COVID-19 patients to one of two arms (1:1 ratio): standard of care or standard of care and very high neutralizing Ab titre convalescent plasma. Randomization will be stratified by centre and by patient cohort. The control group will receive 'standard care' therapy. Neither blinding nor placebo will be used to avoid unnecessary intravenous access.

Standard of care therapy may include anti-SARS-CoV-2 specific medication listed as authorized in the protocol. Centres should ensure that medications used as standard of care are used similarly for patients in both treatment arms.

Participating patients will be included in 2 cohorts of vulnerable patients (cohort 1: elderly (≥ 70 years) and younger with comorbidities (cohort 1: < 70 with comorbidities), cohort 2: immunosuppressed patients).

All subjects will undergo a series of efficacy and safety assessments, including laboratory assays. Subjects will be assessed at baseline, and at Days 3, 14, 28, 90 and 180.

Nasopharyngeal swabs (NP) or lower respiratory tract samples will be obtained at D1 (pre-treatment), and at D3, D14 and D28 (and monthly in case of positivity until of clearance) for cohort 2.

Blood samples will be obtained at D1, D14 and D28 and on the day of hospitalization (if applicable).

The trial is sponsored by the University Hospital of Besançon in France, the German Red Cross in Germany and the NHSBT in the United Kingdom.

ELIGIBILITY:
Cohort 1: Elderly and high COVID-age population:

Inclusion criteria:

* SARS-CoV-2 RNA detected in a specimen, ≤ 7 days after onset of symptoms
* Symptoms of COVID-19 (so including but not limited to: fever; cough; breathlessness; chest pain; wheeze; sore throat; haemoptysis; runny nose; fatigue; muscle or joint pain; confusion; headache; seizures; nausea; vomiting; diarrhoea; abdominal pain; poor appetite; skin ulcers or rash; ear pain; conjunctivitis; anosmia; bleeding; lymphadenopathy. The attending clinician will determine if symptoms are consistent with COVID-19.
* Clinical status not requiring admission to hospital for COVID-19 disease and oxygen support
* Ability to transfuse (per randomisation) within 7 days after onset of symptoms
* Men or women, 70 years or older OR
* under 70 years with significant comorbidities (arterial hypertension, diabetes, obesity, asthma or other chronic pulmonary disease, cardiovascular disease, cerebrovascular disease, chronic kidney disease / dialysis, hemoglobinopathies, liver disease, chronic neurological disease, rheumatoid arthritis, lupus or psoriasis) resulting in a 'COVID-age' of 70 years or more according to the ALAMA risk calculator https://alama.org.uk/covid-19-medical-risk-assessment/

Exclusion Criteria:

* Age < 18 years (France and Germany only)
* Prior or concurrent treatment for COVID-19 (unless listed as authorized)
* History of COVID-19 disease in the last 90 days prior to enrollment
* Prior anti-SARS-CoV-2 immunization
* Contraindication to receiving CCP including previous history of transfusion-related acute lung injury (TRALI) or moderate or severe allergic reaction to blood components
* Known participant objection to receiving plasma products
* Primary or acquired immune deficiency listed below (see cohort 2)
* Refusal to participate expressed by patient or legally authorised representative
* Pregnancy

Cohort 2: High-risk immunocompromised population

Inclusion criteria:

* SARS-CoV-2 RNA, or positive antigenic test, detected in a specimen, ≤ 7 days after onset of symptoms
* Symptoms of COVID-19 (so including but not limited to: fever; cough; breathlessness; chest pain; wheeze; sore throat; haemoptysis; runny nose; fatigue; muscle or joint pain; confusion; headache; seizures; nausea; vomiting; diarrhoea; abdominal pain; poor appetite; skin ulcers or rash; ear pain; conjunctivitis; anosmia; bleeding; lymphadenopathy. The attending clinician will determine if symptoms are consistent with COVID-19.
* Clinical status not requiring admission to hospital for COVID-19 disease and oxygen support
* Ability to transfuse (per randomisation) within 7 days after onset of symptoms
* Male or female with extremely high risk including:

  a. Patients with at least one of the following acquired immune deficiencies

  i. Lymphoid malignancies treated within the last 12 months ii. Lymphoid malignancies with persistent hypogammaglobulinaemia (IgG < 5g/L) iii. Myeloid malignancies treated by chemotherapy within the last 12 months iv. Myeloid malignancies treated by anti-BCL-2 drugs within the last 12 months v. Myeloid malignancies associated with prolonged neutropenia (≥ 6 weeks) vi. Solid tumour undergoing treatment with chemotherapy (until 3 months after completion of the last chemotherapy cycle) vii. Allogenic hematopoietic stem cell transplantation within the last 12 months or anytime if on-going treatment for chronic GVHD viii. Organ transplantation ix. Anti-B (CD20/CD19) MoAb and/or mycophenolate mofetil treatment within the last 12 months x. Anti-CD19/CD20 CAR-T cell treatment xi. ATG or alemtuzumab treatment within the last 6 months xii. AIDS

OR b. Patients with primary lymphoid immune deficiencies. i. B cell deficiencies (such as Bruton agammaglobulinemia) ii. T cell deficiencies (such as Wiskott Aldrich disease) iii. Combined deficiencies (such as Common variable immunodeficiency).

OR c. Patients without detectable seroconversion ≥ 3 weeks after complete vaccination schedule with an approved vaccine.

Exclusion Criteria:

* Age < 18 years (France and Germany only)
* Prior or concurrent treatment for COVID-19 (dexamethasone, anti-IL-6/IL6R, remdesivir) except for prophylactic administration of anti-SARS-CoV-2 monoclonal antibodies (pre or post exposure) and authorized specific treatment
* History of COVID-19 disease in the last 90 days prior to enrollment
* Contraindication to receiving CCP including previous history of transfusion-related acute lung injury (TRALI) or moderate or severe allergic reaction to blood components
* Known participant objection to receiving plasma products
* Refusal to participate expressed by patient or legally authorised representative
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with hospitalisation with progressive COVID-19 symptoms or death | Day 28
  Proportion of participants with (1) at least one overnight stay in hospital for progressive COVID-19 symptoms or (2) who died

SECONDARY OUTCOMES:
Proportion of participants with hospitalisation for progressive COVID-19 symptoms or death | Day 14
Proportion of patients with hospitalisation for progressive COVID-19 symptoms requiring O2 support*, or death *O2 support: requirement based on O2 saturation level on room air <=93% or respiration rate >30 | Day 14 and Day 28
All-cause mortality | Day 28, 90, 180
Proportion of patients with supplemental oxygen | Day 14, 28
Proportion of patients with non-invasive ventilation | Day 14, 28
Proportion of patients with intubation and mechanical ventilation | Day 14, 28
Change in 10-point WHO Clinical Progression Scale score | Day 14, 28
  The 10-point WHO clinical progression scale ranges from 0 to 10 (0: uninfected; 10: death)
Duration of hospital admission censored at 28 days | Day 28
Proportion of patients with admission to ITU | Day 14, 28
Duration of ITU admission censored at 28 days | Day 28
Proportion of patients with long COVID-19 symptoms and time to recovery | Day 28, 180
Health-related quality of life assessed by EQ-5D quality of life index | Day 28, 180
  EQ-5D is one of the most widely used Health-related quality of life measure. EQ-5D questionnaires have 5 dimensions: Mobility, Human Autonomy, Current Activities, Pain & Discomfort, "Anxiety & Depression, and all dimensions are described by 5 levels corresponding to patient response choices.
  A quality of life index ranging from less than 0 (worse than death) to 1 (full health) is derived from the answers to the questionnaires.
Number of Serious Adverse Events | 72 hours
  Grade 3/4 adverse events and AE unexpected for their nature, onset, evolution, severity or frequency
Number of Participants with arterial and venous thromboembolic events | Day 28, 90, 180

OTHER OUTCOMES:
Change in SARS-CoV-2 RNA level | Day 3, 14, 28, 180
  Polymerase chain reaction, Cycle Threshold value in oral or nose/throat swab samples at days 3, 14, 28 and 180 after randomisation
Change in anti-SARS-CoV-2 spike antibody levels in blood | Day 14, 28
SARS-CoV-2 whole-genome sequence analysis | Day 1, 28
Proportion and clinical characteristics of patients with cultivable virus | Day 28, 180
Virus sequence variation and cultivability over time, overall and in individuals receiving vs not receiving CCP | Day 1, 28

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Tiberghien, MD, PhD, Study Director — Etablissement Français du Sang, La Plaine Saint-Denis, France; Eric Toussirot, MD, PhD, Principal Investigator — Rheumatology department, CHU Besançon, France; Hubert Schrezenmeier, MD, PhD, Principal Investigator — German Red Cross Blood Transfusion Service Baden-Württemberg-Hessen; Lise Estcourt, MD, PhD, Principal Investigator — NHS Blood and Transplant, Oxford, United Kingdom; David Roberts, MD, PhD, Principal Investigator — NHS Blood and Transplant, Oxford, United Kingdom; Bart Rijnders, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (14):
- CHU Besançon, Besançon, France
- Germany (11):
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen, Baden-Wurttemberg
  - Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg
  - Diakonie-Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg
  - Uniklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Institut für Klinische Transfusionsmedizin (IKT), Ulm, Baden-Wurttemberg
  - Uniklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitätsklinikum Brandenburg, Brandenburg, Brandenburg
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Elblandkliniken Riesa, Riesa, Saxony
  - Charité Medizinische Klinik IV, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
- Erasmus Medical Center, Rotterdam, Netherlands
- NHS Blood and Transplant, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoffmann S, Seidel A, Ludwig C, Vieweg C, Muller R, Hofmann H, Jahrsdorfer B, Wuchter P, Kluter H, Schmidt M, Johnsen M, Burkhardt T, Appl T, Schrezenmeier E, Munch J, Tiberghien P, Schrezenmeier H, Korper S. SARS-CoV-2 convalescent plasma for the controlled clinical trial "COVIC-19": Experience from collection of very high-titer plasma from superimmunized individuals. Transfusion. 2025 Oct;65(10):1888-1902. doi: 10.1111/trf.18394. Epub 2025 Sep 12. PMID 40937925
- [Derived] Hoffmann S, Schrezenmeier E, Desmarets M, Halleck F, Durrbach A, Peters L, Tremmel AT, Seidel A, Fuhrer M, Bachmann F, Schrezenmeier J, Greiner J, Korper S, Hofmann H, Ludwig C, Vieweg C, Jahrsdorfer B, Budde K, Schmidt M, Munch J, Joher N, Daguindau E, Gruner B, Brunotte G, Vauchy C, Seifried E, Bradshaw D, Estcourt LJ, Roberts DJ, Toussirot E, Rijnders B, Tiberghien P, Schrezenmeier H. Early, very high-titre convalescent plasma therapy in clinically vulnerable individuals with mild COVID-19: an international, randomised, open-label trial. EBioMedicine. 2025 Mar;113:105613. doi: 10.1016/j.ebiom.2025.105613. Epub 2025 Feb 27. PMID 40020259
- [Derived] Desmarets M, Hoffmann S, Vauchy C, Rijnders BJA, Toussirot E, Durrbach A, Korper S, Schrezenmeier E, van der Schoot CE, Harvala H, Brunotte G, Appl T, Seifried E, Tiberghien P, Bradshaw D, Roberts DJ, Estcourt LJ, Schrezenmeier H. Early, very high-titre convalescent plasma therapy in clinically vulnerable individuals with mild COVID-19 (COVIC-19): protocol for a randomised, open-label trial. BMJ Open. 2023 Apr 27;13(4):e071277. doi: 10.1136/bmjopen-2022-071277. PMID 37105693